CLINICAL TRIAL: NCT04031885
Title: A Multicenter, Open-Label, Randomized-Controlled Study of Abemaciclib, a CDK4 and 6 Inhibitor, in Combination With Fulvestrant Compared to Chemotherapy in Women With HR Positive, HER2 Negative Metastatic Breast Cancer With Visceral Metastases
Brief Title: A Study of Abemaciclib (LY2835219) in Combination With Fulvestrant Compared to Chemotherapy in Women With HR Positive, HER2 Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision based on the inability to enroll subjects into the trial
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17320; I3Y-MC-JPCU (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2019-07-23; First posted 2019-07-24 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Fulvestrant; Capecitabine; Docetaxel; Taxes; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abemaciclib + Fulvestrant (Experimental): 150 milligram (mg) Abemaciclib given orally twice a day (BID) with 500 mg fulvestrant given by intramuscular (IM) injection on Cycle 1 Day 1 (C1D1) and Cycle 1 Day 15 (C1D15), then Day 1 of each subsequent cycle.
  Interventions: Drug: Abemaciclib; Drug: Fulvestrant
- Standard Chemotherapy (Active Comparator): Standard chemotherapy of physician's choice (capecitabine, docetaxel, nab paclitaxel, or paclitaxel), administered according to product label.
  Interventions: Drug: Standard Chemotherapy

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib + Fulvestrant
Drug: Fulvestrant — Administered IM
  Arms: Abemaciclib + Fulvestrant
Drug: Standard Chemotherapy — Standard chemotherapy of physician's choice administered according to product label.
  Other Names: Capecitabine; Docetaxel; Nab paclitaxel; Paclitaxel
  Arms: Standard Chemotherapy

SUMMARY:
The reason for this study is to compare the efficacy of abemaciclib, in combination with fulvestrant, to that of physician's choice of chemotherapy in women with hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) metastatic breast cancer that has spread to internal organs. Your participation in this trial could last up to 31 months, depending on your cancer type and how you and your tumor respond.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be females of post-menopausal status with HR+, HER2- breast cancer that has spread to internal organs
* Participants must have had at least one endocrine therapy
* Participants must be willing to use a device to answer daily questions about how they are doing for the duration of their participation in the study
* If participant has diarrhea from a previous treatment, they should talk to their doctor to ensure they have recovered enough to participate in this study

Exclusion Criteria:

* Participants must not have breast cancer that has spread to the brain if untreated and with symptoms
* Participants must not have had any systemic treatment after their breast cancer has spread unless it is endocrine therapy
* Participants must not have certain active infections including HIV or hepatitis
* Participants must not be pregnant or breastfeeding
* Participants must not have certain types of cancers or certain previous cancer treatments
* Participants must not have certain serious medical conditions, including heart or lung disease, or have had certain types of tissue or organ transplants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (61):
- United States (55):
  - Scottsdale Healthcare Hospitals, Avondale, Arizona
  - University of Arizona Cancer Center, Phoenix, Arizona
  - Yuma Regional Cancer Center, Yuma, Arizona
  - CARTI Cancer Center, Little Rock, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Compassionate Cancer Care Medical Group Inc, Corona, California
  - Chan Soon- Shiong Institute for Medicine, Costa Mesa, California
  - Chan Soon- Shiong Institute for Medicine, El Segundo, California
  - Compassionate Cancer Care Medical Group Inc, Fountain Valley, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Scripps Clinic, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - TRIO - Translational Research in Oncology-US, Inc., Los Angeles, California
  - Univ of California Irvine College of Medicine, Orange, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Emad Ibrahim, MD, INC, Redlands, California
  - Compassionate Cancer Care Medical Group Inc, Riverside, California
  - University of California, Davis - Health Systems, Sacramento, California
  - Torrance Memorial Medical Center, Torrance, California
  - Banner MD Anderson Cancer Center, Greeley, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Millennium Oncology, Hollywood, Florida
  - Ocala Oncology, P.A., Ocala, Florida
  - Tallahassee Memorial Cancer Center, Tallahassee, Florida
  - Cleveland Clinic of Florida, Weston, Florida
  - Candler Medical Oncology Practice, Savannah, Georgia
  - Tift Regional Health System Anita Stewart Oncology Center, Tifton, Georgia
  - Kaiser Permanente Center for Health Research, Honolulu, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Cancer Center of Kansas, Wichita, Kansas
  - Touro Infirmary, New Orleans, Louisiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - York Hospital, York Village, Maine
  - Reliant Medical Group, Inc., Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Baptist Cancer Center, Oxford, Mississippi
  - St. Francis Medical Center, Grand Island, Nebraska
  - Oncology Hematology West, Omaha, Nebraska
  - OptumCare Cancer Care, Las Vegas, Nevada
  - Carol Simon Cancer Center at Overlook Medical Center, Summit, New Jersey
  - Brooklyn Methodist Hospital, Brooklyn, New York
  - Weill Cornell Medical College, New York, New York
  - SUNY At Stony Brook, Stony Brook, New York
  - White Plains Hospital, White Plains, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cancer Care Associates of York, York, Pennsylvania
  - Womens and Infants, Providence, Rhode Island
  - Baptist Cancer Center, Memphis, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Providence Regional Cancer Partnership, Everett, Washington
  - Cancer Care Northwest, Spokane, Washington
- Puerto Rico (6):
  - Centro Integrado de Cancer del Sur, PSC, Coto Laurel, PR
  - Bella Vista Oncology Group, Mayagüez, PR
  - Ponce Medical School, Ponce, PR
  - Centro de Cancer de la Mujer, Ponce, PR
  - Fundacion de Investigacion de Diego, San Juan, PR
  - Clinical Research Puerto Rico, Inc., San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Abemaciclib (LY2835219) in Combination With Fulvestrant Compared to Chemotherapy in Women With HR Positive, HER2 Negative Metastatic Breast Cancer — https://www.lillytrialguide.com/en-US/studies/metastatic-breast-cancer/JPCU#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early as a business decision based on the inability to enroll subjects into the trial.
Pre-assignment Details: Participants who have had at least one adequate tumor assessment at baseline and post-baseline and are off study treatment are considered to have completed the study.
Period: Overall Study
Arm/Group | Abemaciclib + Fulvestrant | Standard Chemotherapy
Started | 1 | 3
Received Any Quantity of Study Treatment | 1 | 1
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Abemaciclib + Fulvestrant: 150 mg Abemaciclib given orally BID with 500 mg fulvestrant given by IM injection on C1D1 and C1D15, then Day 1 of each subsequent cycle.
- Total: Total of all reporting groups
Arm/Group | Abemaciclib + Fulvestrant | Standard Chemotherapy | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR)
Description: ORR is defined as the number of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the total number of participants randomized to the corresponding treatment arm [intent-to-treat (ITT) population], based on investigator-assessed tumor responses.CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking in reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. Confirmations of CR and PR are not required.
Time Frame: Randomization to Measured Progressive Disease (Up to 12 Months)
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- Abemaciclib + Fulvestrant: 150 mg Abemaciclib given orally BID with 500 mg fulvestrant given by IM injection C1D1 and C1D15, then Day 1 of each subsequent cycle.
Arm/Group | Abemaciclib + Fulvestrant | Standard Chemotherapy
Number analyzed (Participants) | 1 | 3
percentage of participants | 0 | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from first dose date until the first occurrence of documented disease progression per Response Criteria In Solid Tumors version 1.1(RECIST v1.1) or death from any cause in the absence of progressive disease. Progression-free survival will be based on investigator-assessed tumor responses; there will not be an independent central review of imaging data.
Time Frame: First Dose Date to Objective Progression or Death Due to Any Cause (Up to 12 Months)
Population: Zero participants analyzed, no data collected.
Arm/Group | Abemaciclib + Fulvestrant | Standard Chemotherapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from first dose date until the date that measurement criteria for CR or PR (whichever is first recorded) are first met, per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: First Dose to Date of CR or PR (Up to 12 Months)
Population: Zero participants analyzed, no data collected.
Arm/Group | Abemaciclib + Fulvestrant | Standard Chemotherapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date that measurement criteria for CR or PR (whichever is first recorded) are first met until the first date that disease is recurrent or documented disease progression is observed, per RECIST 1.1 criteria, or the date of death from any cause in the absence of documented disease progression or recurrence.
Time Frame: Date of CR or PR to Date of Objective Progression or Death Due to Any Cause (Up to 12 Months)
Population: Zero participants analyzed, no data collected.
Arm/Group | Abemaciclib + Fulvestrant | Standard Chemotherapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression Free Survival 2 (PFS 2)
Description: PFS 2 is defined as the time from first dose date to the disease progression date on next line (first line of post-discontinuation treatment), or starting date of the second line of post-discontinuation treatment or death from any cause, whichever is earlier, or death from any cause, whichever is earlier.
Time Frame: Randomization to Second Objective Progression or Death Due to Any Cause (Up to 12 Months)
Population: Zero participants analyzed, no data collected.
Arm/Group | Abemaciclib + Fulvestrant | Standard Chemotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 12 months
Description: All randomized participants who received any quantity of study treatment.
Arm/Group | Abemaciclib + Fulvestrant | Standard Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + Fulvestrant (N=1) | Standard Chemotherapy (N=3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + Fulvestrant (N=1) | Standard Chemotherapy (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (2)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Mucosal pigmentation (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (4)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (6)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early as a business decision based on the inability to enroll subjects into the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT04031885/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT04031885/SAP_001.pdf